CLINICAL TRIAL: NCT00264979
Title: Prospective Randomized Study Comparing the Morbidity and Mortality After Liver Resection for Synchronous Colorectal Cancer Metastases When Performed Either During or 12 to 14 Weeks After the Primary Resection
Brief Title: Evaluation of 2 Resection Strategies of Synchronous Colorectal Cancer Metastases
Acronym: METASYNC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stop recommended following the last sequential analysis
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGS 2005/0193; PHRC/04-01; CIC0203/030
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer; Hepatic Metastases
Keywords: Colorectal cancer; Sequential or simultaneous surgery; Synchronous hepatic metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Overlapping Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Simultaneous surgery of colorectal cancer and synchronous liver metastases
  Interventions: Procedure: Simultaneous surgery
- 2 (Other): Sequential surgeries of colorectal cancer and synchronous liver metastases
  Interventions: Procedure: Sequential surgery

INTERVENTIONS:
Procedure: Simultaneous surgery — Simultaneous surgery of colorectal cancer and synchronous liver metastases
  Arms: 1
Procedure: Sequential surgery — Sequential surgeries of colorectal cancer and synchronous liver metastases: the metastases surgery will be programmed 12 to 14 weeks after the primary tumour exeresis.
  Arms: 2

SUMMARY:
The surgical strategy for the treatment of synchronous colorectal cancer liver metastases has not still been defined. The purpose of this study is to compare two treatment strategies in which liver resection is performed either during, or 12 to 14 weeks after the primary resection. Endpoints include the rate of severe complications and survival.

DETAILED DESCRIPTION:
In France, 35 000 colorectal cancers are diagnosed each year, 15 to 25% of which with hepatic metastases. It is nowadays admitted that the complete resection of these hepatic metastases represents the only treatment that has been shown to increase survival. The aim of this study is to evaluate the efficacy/safety ratio of the liver surgery when performed simultaneously or at distance of the primitive tumour ablation. Patients are randomized to undergo liver surgery either during, or 12 to 14 weeks after the primary resection. The primary endpoint is the rate of patients with at least one severe complication within 60 days after surgery. Secondary endpoints evaluate long-term clinical outcomes, in particular recurrence-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults over 18 years old
* At least one adenocarcinoma of colon and/or rectum, histologically proven.
* No local complication at the time of surgery (no occlusion, no sub-occlusion, no massive hemorrhage, no abscesses or local invasion)
* At least one hepatic metastasis which R0 resection is possible through a conventional simple resection
* Informed written consent.

Non inclusion criteria:

* Heart, Respiratory or Renal failure
* Physical or psychological dependence
* Chronic liver disease
* Extra-hepatic metastases

Exclusion Criteria (at time of surgery)

* Localized or diffuse peritoneal carcinomatosis
* Non resectable lymph node metastases
* Colorectal or hepatic tumour extension towards abdominal wall and/or adjacent organ making liver R0 resection impossible immediately
* Other hepatic lesions diagnosed with ultrasound making liver R0 resection impossible immediately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-03-02 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Rate of patients with at least one postoperative severe complication within 60 days after each surgery | 60 days after each surgery

SECONDARY OUTCOMES:
Death rate during hospitalization or within 60 days after each surgery | 60 days after each surgery
Rate and number of severe general, digestive or hepatic complications | 2 years after the first surgery
Rate of unachieved hepatic resection | Day of the hepatic surgery
Global survival distribution and 2 years global survival rate | 2 years after the first surgery
Recurrence-free survival distribution and 2 years recurrence-free survival rate | 2 years
Two years recurrence rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karim Boudjema, MD, PhD, Principal Investigator — CHU Rennes; Jean-Luc Raoul, MD, Principal Investigator — Centre Eugène Marquis - CRLCC Rennes; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes
Locations (14):
- France (14):
  - Chirurgie générale viscérale et digestive - Hôpital Nord, Amiens
  - Service de Chirurgie viscérale, digestive et cancérologie - Hôpital Jean Mingoz, Besançon
  - Chirurgie digestive, thoracique et cancérologie, Dijon
  - Département de Chirurgie - CRLCC Léon Bérard, Lyon
  - Clinique Chirurgicale A - Hôtel Dieu, Nantes
  - Clinique Chirurgicale I - Hôpital Nord, Nantes
  - Centre de Chirurgie et Réanimation Digestives - Hôpital Saint Antoine, Paris
  - Service de Chirurgie hépato-biliaire et Transplantation Hépatique- Paris Saint Antoine, Paris
  - Service de Chirurgie - Hôpital Jean Bernard, Poitiers
  - Service d'Oncologie Digestive- CRLCC Eugène Marquis, Rennes
  - Département de Chirurgie Viscérale - Hôpital Pontchaillou, Rennes
  - Centre de Chirurgie Viscérale et de Transplantation - CHU de Hautepierre, Strasbourg
  - Chirurgie Viscérale Digestive - CH Chubert, Vannes
  - Centre Hépato-biliaire - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Background] Martin R, Paty P, Fong Y, Grace A, Cohen A, DeMatteo R, Jarnagin W, Blumgart L. Simultaneous liver and colorectal resections are safe for synchronous colorectal liver metastasis. J Am Coll Surg. 2003 Aug;197(2):233-41; discussion 241-2. doi: 10.1016/S1072-7515(03)00390-9. PMID 12892803
- [Background] Weber JC, Bachellier P, Oussoultzoglou E, Jaeck D. Simultaneous resection of colorectal primary tumour and synchronous liver metastases. Br J Surg. 2003 Aug;90(8):956-62. doi: 10.1002/bjs.4132. PMID 12905548